CLINICAL TRIAL: NCT03085173
Title: A Phase I Trial of CD19-Targeted EGFRt/19-28z/4-1BBL "Armored" Chimeric Antigen Receptor (CAR) Modified T Cells in Patients With Relapsed or Refractory CD19+ Hematologic Malignancies
Brief Title: A Trial of "Armored" CAR T Cells Targeting CD19 For Patients With Relapsed CD19+ Hematologic Malignancies
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Juno Therapeutics, Inc., a Bristol-Myers Squibb Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-1570
Record Dates: First submitted 2017-03-15; First posted 2017-03-21 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-04

CONDITIONS: Chronic Lymphocytic Leukemia (CLL); Relapsed; Refractory
Keywords: CAR T Cells Targeting CD19; EGFRt/19-28z/4-1BBL; 16-1570
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Recurrence

STUDY DESIGN:
Intervention Model Description: A Phase I Trial of CD19-Targeted EGFRt/19-28z/4-1BBL "Armored" Chimeric Antigen Receptor (CAR) Modified T Cells in Patients with Relapsed or Refractory Chronic Lymphocytic Leukemia (CLL)
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- EGFRt/19-28z/4-1BBL CAR T cells (Experimental): Following enrollment, patients will undergo leukapheresis of peripheral blood for further T cell enrichment, activation and genetic modification using a retroviral vector encoding a CD19targeted CAR, the co-stimulatory ligand 4-1BBL and the EGFRt safety system (EGFRt/19-28z/4-1BBL). These T cells will be expanded and after the appropriate number of cells is generated, the modified T cells may be infused fresh or frozen for later use according to standard operation procedures. Modified T cell infusions will be administered 2-7 days following completion of the treating investigator's choice of conditioning chemotherapy. Serial sampling of blood and bone marrow will be performed following treatment to assess toxicity, therapeutic effects, and survival of the genetically modified T cells.
  Interventions: Biological: EGFRt/19-28z/4-1BBL CAR T cells

INTERVENTIONS:
Biological: EGFRt/19-28z/4-1BBL CAR T cells — Cohorts of 3-6 patients will be infused with escalating doses of EGFRt/19-28z/4-1BBL CAR T cells to establish the maximum tolerated dose (MTD). There are 4 planned dose levels: 1 x 10^5, 3 x 10^5, 1 x 10^6, and 3 x 10^6 CAR T cells/kg.

SUMMARY:
The purpose of this phase I study is to test the safety of different dose levels of specially prepared cells collected from the patient called "modified T cells". The investigators want to find a safe dose of modified T cells for patients with this type of cancer that has progressed after standard therapy. The investigators also want to find out what effects these modified T cells have on the patient and the cancer.

For patients who were treated, had progression of disease and were removed from study, duplicate enrollment is permitted if it is determined the patients could receive a benefit. If the patients meet all eligibility criteria, they can be enrolled onto study a second time as a new accrual, and receive treatment in a higher dose level cohort.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have CD19+ B cell malignancy with relapsed or refractory disease, defined as below:

Patients with CLL:

* Refractory to or relapsed after at least 2 prior chemo or chemoimmunotherapy (e.g. FCR, BR) requiring further treatment
* Refactory to or relapsed after at least 1 prior biologic agent (e.g. Ibrutinib, idelalisib, venetoclax, except a single agent anti-CD20 monoclonal antibody) requiring further treatment

Patients with iNHL (FZ, MZL, WM):

* Refractory or relapsed after at least 2 lines of chemoimmunotherapy (including at least one course of anti-CD20 antibody)
* Refractory or relapsed after at least 1 prior biologic agent (e.g. lenalidomide, ibrutinib, idelalisib)
* Patients must have measurable disease (for WM patients, measureable disease is demonstrable monoclonal paraprotein and bone marrow involvement)

Patients with DLBCL, Transformed B cell lymphoma, or High grade B cell lymphoma:

* Refractory to or relapsed after 1 or more prior chemoimmunotherapies with at least one containing an anthracycline and CD20 directed therapy
* Transplant ineligible
* Biopsy proven relapsed disease

Patients with ALL, CML in lymphoid blast crisis or Burkitt's lymphoma:

* Refractory to at least 1 prior induction chemotherapy
* Relapsed after at least 1 prior multiagent systemic chemotherapy that included induction and consolidation
* Patients with Philadelphia chromosome-positive ALL must have failed a second generation tyrosine kinase inhibitor

  * Age ≥ 18 years of age
  * Creatinine ≤2.0 mg/100 ml, direct bilirubin ≤2.0 mg/100 ml, AST and ALT ≤3.0x upper limit of normal (ULN)
  * Adequate pulmonary function as assessed by ≥92% oxygen saturation on room air by pulse oximetry

Exclusion Criteria:

* Karnofsky performance status <70
* Pregnant or lactating women. Women and men of childbearing age should use effective contraception while on this study and continue for 1 year after all treatment is finished
* Impaired cardiac function (LVEF <40%) as assessed by ECHO or MUGA scan
* Patients with active known autoimmune disease are ineligible
* Patients with following cardiac conditions will be excluded:

  * New York Heart Association (NYHA) stage III or IV congestive heart failure
  * Myocardial infarction </= 6 months prior to enrollment
  * History of clinically significant ventricular arrhythmia or unexplained syncope, not believed to be vasovagal in nature or due to dehydration <6 months prior to enrollment
  * History of severe non-ischemic cardiomyopathy with EF </=20%
* Patients with HIV or active hepatitis B or hepatitis C infection are ineligible
* Patients with uncontrolled systemic fungal, bacterial, viral or other infection are ineligible
* Patients with any concurrent active malignancies as defined by malignancies requiring any therapy other than expectant observation or hormonal therapy, with the exception of squamous and basal cell carcinoma of skin
* Patients with history or presence of clinically significant neurological disorders such as epilepsy, generalized seizure disorder, severe brain injuries are ineligible
* Any other issue which, in the opinion of the treating physician, would make the patient ineligible for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | occurring within 30 days from the last infusion
  Cohorts of 3-6 patients each will be treated with escalating doses of modified T cell. At least 3 patients will be treated at each dose level with an accrual of no more than 2 patients per month within each dose level. At least two weeks will elapse from the first patient's T cell infusions before the second patient is treated (on dose level 1) to allow for toxicity and safely assessment. All patients treated at the preceding dose level will be observed a minimum of 4 weeks before dose escalation occurs.

CONTACTS AND LOCATIONS:
Overall Officials: Jae Park, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm